CLINICAL TRIAL: NCT00559416
Title: Immunologic and Virologic Response in HIV Infected Progressors After Infusion of Lymphocytes From HIV Infected "Elite" Long-Term Non-Progressors
Brief Title: Lymphocyte Infusions for the Treatment of HIV-Infected Patients Failing Anti-HIV Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080024; 08-CC-0024
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2016-09-30

CONDITIONS: HIV Infections
Keywords: HIV/AIDS; HLA-B*57; Cell Transfer; HIV; treatment experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Drug: Cell Transfer

SUMMARY:
Some HIV-infected individuals have a white blood cell marker known as HLA-B*57 that appears to help control the progress of the disease; however, not all who have the HLA-B*57 marker are able to control the infection. This study will examine the effects of giving white blood cells with HLA-B*57 from an individual who controls HIV infection to an individual who cannot control HIV infection, as a form of HIV treatment. All candidates will be screened with a medical history, physical examination, and blood and urine tests.

Both donor and recipient volunteers must be HIV-positive individuals 18 years of age or older who have the HLA-B*57 marker and are receiving care. Donor candidates must have positive HIV antibody tests for at least seven years with a recent CD4 cell count greater than 400 cells/mm?, HIV viral load less than 50 copies/mL, and no previous HIV viral load greater than 1,000 copies/mL. Recipient candidates must have positive HIV antibody tests with a recent CD4 cell count less than 400 cells/mm? and HIV viral load greater than 10,000 copies/mL, and must have failed at least two prior combination antiretroviral regimes and are willing to receive or resume combination antiretroviral therapy. Donor volunteers will be excluded if they have taken certain antiretrovirals drugs, have a medical history of cancer or of other blood-borne illnesses, or have other medical conditions that might interfere with the study. Recipient volunteers will be excluded if they have a medical history of malignant cancer or other medical conditions that might possibly interfere with the study.

Donors will undergo apheresis to separate white blood cells from circulating blood before the red blood cells and plasma are returned to the bloodstream. The procedure will take up to five hours, and donors will be required to return for additional tests. Donors may be asked to return for further white blood cell donations, a maximum of six procedures per year.

Recipients will undergo apheresis to obtain stem cells for possible use in the study, and will be admitted to an NIH Clinical Center inpatient unit to receive an infusion of white blood cells and undergo a series of blood tests both before and after the infusion. The infusion process will take two hours. After being discharged, recipients will be asked to return to the Clinical Center for monitoring and follow-up tests, and may receive further infusions.

DETAILED DESCRIPTION:
Improvements in human immunodeficiency virus/acquired immunodeficiency syndrome (HIV/AIDS) treatments in the United States have made the disease in many cases a chronic illness. However, many individuals have failed multiple lines of standard therapy, and thus, development of new modes of salvage treatment is crucial. Restriction of viral replication, mediated by CD8+ cells, appears to play an important role in control of HIV replication. A subset of individuals, many of whom possess human leukocyte antigen (HLA) B*57 exhibit restriction of HIV type 1 viral replication to less than 50 copies/mL, presumably by a mechanism that is CD8+ T-cell mediated, and become elite long-term non-progressors (LTNP), who have no evidence of progressive immunodeficiency and no development of opportunistic complications during many years of follow-up. Other individuals, including those with HLA-B*57 show no evidence of control of HIV replication, and without antiretroviral therapy will develop progressive immunodeficiency and HIV-related opportunistic complications. In this exploratory study, we are investigating a novel cell transfer strategy: up to 3 patients with HIV infection have failed at least 2 standard regimens of antiretroviral therapy, have a CD4+ count under 200 cells/mm (3), and a plasma HIV viral load of greater than 10,000 copies/mL, will be administered 10 (10) peripheral blood mononuclear cells obtained by lymphapheresis from an "elite" LTNP matched to the recipient on at least one HLA-B allele. Up to 70 patients may be enrolled for screening to identify 3 donors and 3 recipients. Up to 3 infusions may be administered per patient, with each infusion occurring no more frequently than every 3 months. The primary endpoints will be the safety of the infusions and the survival of donor cells in the recipient. Changes in the recipient s CD4+ and CD8+ cell number, other immune parameters, and plasma HIV viral load will also be monitored closely for evidence of anti-HIV activity.

ELIGIBILITY:
* INCLUSION CRITERIA RECIPIENT:

Under this protocol, cell recipients must fulfill all of the following characteristics and conditions:

Greater than or equal to 18 years old

Ability to sign informed consent

For women of child-bearing potential, negative result on a serum or urine pregnancy test; in addition, men and women of childbearing potential must agree to practice abstinence or use two methods of birth control/contraception (condoms, diaphragm or cervical cap with spermicide, IUD, or hormonal-based contraception) for at least 4 weeks after each cell infusion

Willingness to comply with study requirements and procedures including storage of blood for possible future use to study HIV/AIDS, related diseases, or the immune system

Willingness to permit HLA testing

Hematocrit greater than or equal to 27 percent, platelets greater than or equal to 25,000/mm (3)

No significant underlying cardiac, renal, or hepatic disease (Creatinine less than 2.0 mg/dL; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 150 U/mL)

HIV infection must be confirmed by ELISA and a confirmatory test (e.g. western blot if not previously documented, and patients must be under the care of a primary care physician.

Viral load greater than 10,000 copies/mL on available optimized combination antiretroviral therapy, to include at least 3 drugs, one of which is a non-nucleoside reverse transcriptase inhibitor (NNRTI), integrase inhibitor, or protease inhibitor. Patients not on combination antiretroviral therapy will be eligible, but must be willing to resume combination antiretroviral therapy and to have had a viral load greater than 10,000 copies/mL after at least 2 weeks of therapy.

Failure or intolerance of at least two previous combination antiretroviral regimens. Failure will be defined as an HIV viral load greater than 400 copies/mL while taking a given regimen.

Recipient must be taking appropriate prophylaxis for opportunistic infections, as per Public Health Service (PHS) guidelines, unless there is intolerance to available medications.

Screening CD4+ cell count less than or equal to 350 cells/mm(3) obtained within 6 weeks prior to study entry.

EXCLUSION CRITERIA FOR RECIPIENT:

An individual will be ineligible to receive cells if one or more of the following conditions are present:

Discordance with donor on antibody status of EBV, CMV, or HHV-8 if donor is antibody positive for EBV, CMV, or HHV-8.

Malignancy requiring systemic therapy, or a history of malignancy that required myelotoxic chemotherapy.

Active untreated opportunistic infection that requires systemic therapy. Patients with opportunistic infections who have received greater than 2 weeks of therapy will be eligible.

Is pregnant or breast feeding.

Severe psychiatric disorder that would interfere with adherence to protocol requirements. Individuals who have a stable psychiatric condition may be eligible.

Current use or a history of treatment with investigational agent(s) within 3 months of protocol enrollment. ARVs obtained through expanded access programs are permitted.

Current use or a history of treatment with a systemic corticosteroid, immunosuppressive, or cytotoxic agent within 30 days of protocol enrollment.

Any other medical condition for which the investigator believes cell transfer may be contraindicated.

Ever been diagnosed with autoimmune vasculitis.

INCLUSION CRITERIA DONOR:

Donor eligibility criteria as specified by the FDA will be followed, except for HIV testing. All donors will be HIV positive as per protocol and as described in the IND application. Under this protocol, cell donors must fulfill all of the following characteristics and conditions:

Greater than or equal to 18 years old.

Ability to sign informed consent.

For women of child-bearing potential, negative result on a serum or urine pregnancy test.

Willingness to comply with study requirements and procedures including storage of blood for possible future use to study HIV/AIDS, related diseases, or the immune system.

Willingness to permit HLA testing.

Matched to at least one HLA-B allele of the potential recipient. The

match will be at a two-digit resolution HLA allele level of typing or higher.

Hematocrit greater than or equal to 30 percent, platelets greater than or equal to 100,000/mm(3), white blood cells greater than or equal to 3.0 times 10(9)/L.

No underlying cardiac, pulmonary, renal, or hepatic disease that would preclude patient from undergoing apheresis.

HIV infection must be confirmed by ELISA and a confirmatory test (e.g. western blot if not previously on record, and patients must be under the care of a primary care physician.

HIV infection for greater trhan or equal to 7 years.

For patients with a history of no or minimal (one or two nucleotide reverse transcriptase inhibitor (NRTI) drugs) prior antiretroviral therapy: CD4+ cell count greater than or equal to 400 cells/mm(3) and HIV viral load less than 50 copies/mL, with no recorded HIV viral load obtained after acute HIV infection greater than 2,500 copies/mL. For patients currently receiving antiretroviral therapy: no antiretroviral therapy for a period of at least 7 years prior to starting antiretroviral therapy, with CD4+ cell count greater than or equal to 400 cells/mm(3) and HIV viral load < 50 copies/mL at the time of initiation of antiretroviral therapy, and no recorded HIV viral load obtained after acute HIV infection > 2,500 copies/mL. HIV viral loads obtained during acute HIV infection (within 6 months of the estimated date of seroconversion) will not be utilized for study inclusion/exclusion.

Minimum wt of 110 lbs<TAB>

EXCLUSION CRITERIA FOR DONOR:

An individual will be ineligible to donate cells if one or more of the following conditions are present:

Ever having been diagnosed with any AIDS-defining illnesses

Positive results on screening test for any of the following tests: HCV enzyme immunoassay (EIA) repeat reactive/ recombinant immunoblot (RIBA) confirmed, HBV/HCV NAT, HTLV-I/II antibodies, T.cruzi antibodies, HBsAg, or serologic test for syphilis (with positive confirmatory treponemal-based assay), unless the patient has received adequate therapy for syphilis. Donors with a positive West Nile Virus NAT are deferred for 120 days.

Is pregnant or breast feeding

HLA homozygous donor who is haplo-identical to recipient

History of malignancy other than basal cell carcinoma of the skin, or in situ carcinoma of cervix or colon

ALT or AST greater than 2 times the upper limit of normal

Been diagnosed with malaria

Been diagnosed with Chagas disease

Been diagnosed with babesiosis

Received a dura mater (or brain covering) graft

Been diagnosed with any neurological disease

Relative had Creutzfeldt-Jakob disease

Had a transplant or other medical procedure that involved being exposed to live cells, tissues, or organs from an animal

Had a sexual partner or a member of the household have a transplant or other medical procedure that involved being exposed to live cells, tissues, or organs from an animal

Severe psychiatric disorder that would interfere with adherence to protocol requirements. Individuals who have a stable psychiatric condition may be eligible.

Current use or a history of treatment with investigational agent(s) within 3 months of protocol enrollment.

Current use or a history of treatment with a systemic corticosteroid, immunosuppressive, or cytotoxic agent within 30 days of protocol enrollment.

Any other medical condition for which the investigator believes apheresis may be contraindicated.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-11-08; Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Safety, survival of transferred cells.

SECONDARY OUTCOMES:
Changes in immune and viral parameters (CD4, Plasma HIV levels)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Kovacs, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Coffin JM. HIV population dynamics in vivo: implications for genetic variation, pathogenesis, and therapy. Science. 1995 Jan 27;267(5197):483-9. doi: 10.1126/science.7824947.
- [Background] Rosenberg ES, Billingsley JM, Caliendo AM, Boswell SL, Sax PE, Kalams SA, Walker BD. Vigorous HIV-1-specific CD4+ T cell responses associated with control of viremia. Science. 1997 Nov 21;278(5342):1447-50. doi: 10.1126/science.278.5342.1447. PMID 9367954
- [Background] Kovacs JA, Lempicki RA, Sidorov IA, Adelsberger JW, Sereti I, Sachau W, Kelly G, Metcalf JA, Davey RT Jr, Falloon J, Polis MA, Tavel J, Stevens R, Lambert L, Hosack DA, Bosche M, Issaq HJ, Fox SD, Leitman S, Baseler MW, Masur H, Di Mascio M, Dimitrov DS, Lane HC. Induction of prolonged survival of CD4+ T lymphocytes by intermittent IL-2 therapy in HIV-infected patients. J Clin Invest. 2005 Aug;115(8):2139-48. doi: 10.1172/JCI23196. Epub 2005 Jul 14. PMID 16025158
- [Derived] Migueles SA, Chairez C, Lin S, Gavil NV, Rosenthal DM, Pooran M, Natarajan V, Rupert A, Dewar R, Rehman T, Sherman BT, Adelsberger J, Leitman SF, Stroncek D, Morse CG, Connors M, Lane HC, Kovacs JA. Adoptive lymphocyte transfer to an HIV-infected progressor from an elite controller. JCI Insight. 2019 Sep 19;4(18):e130664. doi: 10.1172/jci.insight.130664. PMID 31415245